CLINICAL TRIAL: NCT05391438
Title: Impact of Meal Timing on Glycemic Profile in Latino Adolescents With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Alaina P. Vidmar, MD, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHLA-22-00119
Record Dates: First submitted 2022-05-19; First posted 2022-05-26 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Obesity; Meal Timing
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: proof-of-concept study to measure glycemic and metabolic responses to a test meal (controlled for macronutrient profile and caloric amount) administered at various times of the day (early vs. afternoon vs. late) in thirty Latino adolescents. All participants will consume three standard test meals administered in random order at different times of day over two-weeks: (1) Early: test meal consumed at 8 AM; (2) Afternoon: test meal consumed at 12 PM; (3) Late: test meal consumed at 4 PM. A continuous glucose monitor (CGM) will be placed on the participant for the duration of the 2-week period. Baseline and post-meal samples will be assayed for glucose, insulin, c-peptide, GLP-1, GIP, PP at times -10, -5, 0, 10, 20, 30, 45, 60, 90, 120, 150 and 180 minutes after glucose. The primary endpoints will be glucose, insulin, and C-peptide area under the curve, insulinogenic index, and glucose variability as captured by percent time in range on CGM following the test meal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meal-timing (Other): All participants will consume three standard test meals administered in random order at different times of day over two-weeks: (1) Early: test meal consumed at 8 AM; (2) Afternoon: test meal consumed at 12 PM; (3) Late: test meal consumed at 4 PM. A continuous glucose monitor (CGM) will be placed on the participant for the duration of the 2-week period.
  Interventions: Other: Meal-timing

INTERVENTIONS:
Other: Meal-timing — We propose a cross-over, proof-of-concept study to measure glycemic and metabolic responses to a test meal (controlled for macronutrient profile and caloric amount) administered at various times of the day (early vs. afternoon vs. late) in thirty Latino adolescents (ages 13-19 years), with obesity, without diabetes, to determine how timing of eating impacts glycemic response to the test meal after a 16-h fasting period. All participants will consume three standard test meals administered in random order at different times of day over two-weeks: (1) Early: test meal consumed at 8 AM; (2) Afternoon: test meal consumed at 12 PM; (3) Late: test meal consumed at 4 PM. A continuous glucose monitor (CGM) will be placed on the participant for the duration of the 2-week period. Baseline and post-meal samples will be assayed for glucose, insulin, c-peptide, GLP-1, GIP, PP at times -10, -5, 0, 10, 20, 30, 45, 60, 90, 120, 150 and 180 minutes after glucose.

SUMMARY:
In adolescents, conventional obesity treatment comprehensively addresses nutritional, activity, and behavioral topics. Due to limited resources in historically marginalized communities, implementation of nutrition-based interventions that require easy access to fresh food and ability to change the home environment is difficult, which may exacerbate health disparities. It is critical to find nutrition strategies and recommendations that are impactful, sustainable, and cost effective across all communities. There is growing interest in time-based interventions focusing on "when" food is consumed rather than on prescribed macronutrient composition. Time-restricted eating (TRE) is a type of meal-timing which involves fasting for at least 14-hours per day and eating over a 10-hour eating window initiated in the morning, mid-day, or afternoon. TRE recommendations are simple in merely dictating when eating occurs and thus may represent a more straightforward approach for adolescents than other caloric restriction regimens relying on numeracy (kilocalories and macronutrients) and goal setting. In adults, early-day TRE has been shown to reduce body weight, fasting glucose, and insulin resistance. By contrast, restricting food intake to the evening has produced mostly null results or even worsened post prandial glucose levels and β-cell responsiveness. To date, there has been no trial comparing early vs. late TRE on glycemic profiles in adolescents, and it is unclear how meal-timing impacts glycemic profiles in youth. The optimal timing of food intake for adolescents may be very different than adults due to increasing sex steroids and growth hormone levels overnight which may contribute to increased insulin resistance in the early morning. The proposed proof-of-concept study addresses this question by measuring metabolic response to a test meal consumed in the morning, afternoon, and evening among 30 adolescents with obesity using a within participant design. These findings will provide the needed research base for the refinement of TRE interventions in adolescence.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes in adolescents is steadily increasing, specifically among Latino youth. Unfortunately, there is a lack of effective preventative treatments available to delay the progression to type 2 diabetes in youth living with obesity and pre-diabetes. Specifically, it is challenging for many adolescents to maintain adherence to multicomponent interventions resulting in high attrition which then decreases efficacy. There is growing interest in time-based interventions focusing on "when" food is consumed rather than on prescribed macronutrient composition. In the adult population there has been increasing evidence that time-restricted eating (TRE), which consists of limiting daily food intake to an 8 to 10-hour period or less may improve insulin sensitivity and β-cell responsiveness. However the results of TRE in adults appear to depend on when eating occurs. Early TRE (last eating event prior to 16:00) has been shown to reduce body weight, fasting glucose and insulin, and insulin resistance. However, restricting food intake to the evening produced mostly null results or worsened post prandial glucose level. One possible explanation is that consuming food early in the day synchronizes the central and peripheral circadian clocks involved in energy expenditure and fat oxidation and minimizes glycemic excursions and endogenous glucose production via enhanced insulin secretion. It has been proposed that the enhanced insulin secretion may be secondary to corresponding diurnal variations in the release of incretin hormones such as glucagon, glucagon-like-peptide-1 (GLP-1), glucose-dependent insulinotropic polypeptide (GIP), and pancreatic peptide (PP).

Because of its simplicity, TRE may represent a more feasible approach for adolescents than other caloric restriction regimens. Our team recently conducted the first study examining the feasibility of TRE in adolescents with obesity. In this study, fifty adolescents were randomized to a self-selected 8-hour TRE compared to a prolonged eating window. TRE was found to be feasible, safe, and acceptable but there was no difference in glycemic profiles or weight loss between groups. These null findings may be due to the late eating window that was selected. To date, there have been no trial comparing early vs. late TRE on glycemic profiles in adolescents and it is unclear how meal-timing impacts glycemic profiles in youth. It remains unknown how the timing of meal consumption directly effects glycemic profiles and cardiometabolic endpoints in this age group. Thus, to address this question, in our proof-of-concept study, the investigators aim to measure glycemic and metabolic responses to a test meal (controlled for macronutrient profile and caloric amount) at various meal-timings (early vs. afternoon vs. late) in thirty Latino adolescents (ages 13-19 years), with obesity, without diabetes. All participants will consume three standard test meals administered in random order at different times of day over a two-week period: (1) Early: test meal consumed at 8 AM; (2) Afternoon: 12 PM; (3) Late: 4 PM. Test meals will be consumed on different days at least three days apart after a minimum of a 16-hour fasting period. A continuous glucose monitor (CGM) will be placed on the participant for the duration of the 2-week period. The primary endpoints will be frequently sampled glucose, insulin, and c-peptide area under the curve (AUC) collected after consumption of a standard test meal, insulinogenic index (IGI: change in insulin/change in glucose over the first 30 min after the load), and glucose variability as captured by percent time in range on CGM. The investigators hypothesize that adolescents with obesity will have reduced AUC and IGI following the later meals compared to the early meal. The investigators will test these hypotheses with the following aims:

Aim 1: Identify how timing of meal consumption after a prolonged 16-h fast affects glucose and insulin response in Latino adolescents with obesity. The investigators will measure insulin secretion, clearance rates, and sensitivity assessed with a) 3-h frequent sampling of glucose, insulin, and c-peptide post meal, b) calculated insulinogenic index, and c) percent time in range measured by CGM. The investigators expect that meal consumption at 12 and 4 PM will be associated with lower post prandial glucose excursions, decreased AUC and IGI, and increased percent time in range compared to that same meal consumed at 8 AM.

Aim 2: Examine the association between timing of meal consumption and incretin and pancreatic hormones in Latino adolescents with obesity. The investigators will collect frequent sampling of glucagon, total GLP-1, GIP, and PP concentrations post-meal to explore how diurnal variation in these hormones impact insulin sensitivity. The investigators expect that meal consumption at 12 and 4 PM will in greater change in incretin and pancreatic hormones concentrations compared to that same meals consumed at 8 AM.

Future Direction: The data collected during this pilot will inform the design of a randomized clinical trial to test the feasibility, safety, and efficacy of early vs. late TRE in adolescents with obesity to reduce glycemic and insulin response for the prevention of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. age 13-19 years
2. Hispanic or Latino defined by the NIH as a person of Cuban, Mexican, Puerto Rican, South or Central American, or other Spanish culture or origin, regardless of race; (3)Tanner stage III and above

(4) body mass index > 95th percentile (5) participant must be willing and able to adhere to the assessments, visit schedules, and eating/fasting periods.

Exclusion Criteria:

1. diagnosis of Prader-Willi Syndrome, brain tumor or hypothalamic obesity
2. serious intellectual disability
3. parent/guardian-reported physical, mental of other inability to participate in the assessments
4. previous bariatric surgery
5. current use of an anti-obesity or other diabetes medication (e.g., phentermine, topiramate, orlistat, GLP-1 agonist, naltrexone, buproprion, or insulin)
6. current participation in other interventional weight loss studies.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alaina Vidmar, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Meal-timing
Started | 22
Completed | 15
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Meal-timing
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.5 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants] — 125 Participants were screened, of which 92 eligible participants were identified, and 22 youth consented to participate in the 14-day trial. Population: 7 subjects withdrew
  Participants
    number analyzed (Participants) | 15
    Female | 3
    Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 22
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulinogenic Index From Baseline After Test Meal From Venous Sample
Description: Baseline and post-meal samples will be assayed for glucose, insulin, and c-peptide at times -10, -5, 0, 10, 20, 30, 45, 60, 90, 120, 150 and 180 minutes after the meal is consumed. The Insulinogenic index (change in insulin/change in glucose over the first 30 min after the load) will be calculated. IGI has been widely used as an index of early phase insulin secretion in clinical studies. It is highly correlated with the acute insulin response on intravenous glucose tolerance test and is considered a reasonable surrogate.
Time Frame: Baseline to Day 14
Measure: Median (Inter-Quartile Range); unit: Microunits per milliliter
Arm/Group | Meal-timing
Number analyzed (Participants) | 15
Microunits per milliliter
  8 AM | 268 [83 to 515]
  12 PM | 215 [111 to 286]
  4 PM | 153 [84 to 266]

2. Primary Outcome: Change in Incremental Glucose Area Under the Curve From Baseline After Test Meal From Venous Sample
Description: Glucose incremental area under curve: The positive area under the post-meal glucose curve after subtracting the glucose value at the start.
Time Frame: Baseline to Day 14
Measure: Median (Inter-Quartile Range); unit: mg/dL·min
Arm/Group | Meal-timing
Number analyzed (Participants) | 15
mg/dL·min
  8 AM | 17705 [15154 to 20152]
  12 PM | 18279 [17614 to 18860]
  4 PM | 19122 [18427 to 20493]

3. Secondary Outcome: Change in Quantifying Glucagon Like Peptide 1 Concentrations From Baseline After Test Meal From Venous Sample
Description: Glucagon like peptide 1 concentrations will be measured in duplicate from plasma samples using Millipore Enzyme-linked Immunosorbent Assays (ELISA) or multiplex assays according to the recommendations of the manufacturer (Birmington, MA).
Time Frame: Baseline to Day 14
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Meal-timing
Number analyzed (Participants) | 15
pg/mL
  8 AM | 6 [1 to 7]
  12 PM | 2 [2 to 10]
  4 PM | 8 [1 to 14]

ADVERSE EVENTS:
Time Frame: 14 days
Groups:
- Early; Afternoon; Late: All participants will consume three standard test meals administered in random order at different times of day over two-weeks: (1) Early: test meal consumed at 8 AM; (2) Afternoon: test meal consumed at 12 PM; (3) Late: test meal consumed at 4 PM. A continuous glucose monitor (CGM) will be placed on the participant for the duration of the 2-week period.
  Meal-timing: We propose a cross-over, proof-of-concept study to measure glycemic and metabolic responses to a test meal (controlled for macronutrient profile and caloric amount) administered at various times of the day (early vs. afternoon vs. late) in thirty Latino adolescents (ages 13-19 years), with obesity, without diabetes, to determine how timing of eating impacts glycemic response to the test meal after a 16-h fasting period. All participants will consume three standard test meals administered in random order at different times of day over two-weeks: (1) Early: test meal consumed at 8 AM; (2) Afternoon: test meal consumed at 12 PM; (3) Late: test meal consumed at 4 PM. A continuous glucose monitor (CGM) will be placed on the participant for the duration of the 2-week period. Baseline and post-meal samples will be assayed for glucose, insulin, c-peptide, GLP-1, GIP, PP at times -10, -5, 0, 10, 20, 30, 45, 60, 90, 120, 150 and 180 minutes after glucose.
Arm/Group | Early | Afternoon | Late
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT05391438/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT05391438/ICF_000.pdf